CLINICAL TRIAL: NCT03502499
Title: Half-normal Saline vs Normal Saline for Irrigation of Open-irrigated Radiofrequency Catheters in Idiopathic Left Ventricular Outflow Tract Arrhythmias Ablation
Brief Title: Half-normal Saline in Idiopathic Left Ventricular Outflow Tract Arrhythmias Ablation
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: slow enrollment
Sponsor: Texas Cardiac Arrhythmia Research Foundation (Other)
Responsible Party: Principal Investigator, Andrea Natale, Executive Medical Director, Texas Cardiac Arrhythmia Research Foundation
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: TCAI_HNS_VA
Record Dates: First submitted 2018-04-04; First posted 2018-04-18 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2022-04

CONDITIONS: Ventricular Arrythmia
MeSH Terms: interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Half-normal saline (Experimental)
  Interventions: Drug: Half-normal saline
- Normal saline (Active Comparator)
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Half-normal saline — Use of half-normal saline as an irrigant for open-irrigated ablation catheters
  Arms: Half-normal saline
Drug: Normal saline — Use of normal saline as an irrigant for open-irrigated ablation catheters
  Arms: Normal saline

SUMMARY:
The study evaluates the use of half-normal saline as an irrigant for open-irrigated catheters during left ventricular outflow tract ventricular arrhythmias ablation. By increasing the efficacy of radiofrequency energy-mediated lesion formation, half-normal saline has the potential to reduce procedural times and improved acute and long-term outcomes.

ELIGIBILITY:
Inclusion criteria

* male or female between 18 and 75 years of age at the time of enrollment
* undergoing first-time radiofrequency ablation for left ventricular outflow tract ventricular arrhythmias
* written informed consent obtained from subject or subject's legal representative and ability for subject to comply with the requirements of the study

Exclusion criteria

* ventricular arrhythmias originating from the right ventricular outflow tract according to the ventricular arrhythmia ECG morphology (i.e., precordial R wave transition at V3 or later)
* ventricular arrhythmias not originating from cardiac outflow tracts
* baseline hyponatremia (serum sodium level < 135 mEq/L)
* pregnant, breastfeeding, or unwilling to practice birth control during participation in the study
* presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the patient or the quality of the data

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-05-16 (Actual); Primary Completion 2022-04 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
total radiofrequency ablation time, and total procedure time | intraprocedural
acute success | intraprocedural
  elimination of the VAs, or <10 morphologically similar PVCs during a 15-minute waiting period
long-term success | 1 year
  elimination of the VAs, or a reduction of >75% of the PVC burden associated with marked improved in symptoms

OTHER OUTCOMES:
procedure-related complications | periprocedural (at the time of the procedure and up to 1 month)
  pericardial effusion due to cardiac perforation or pericarditis, transient ischemic attack/stroke, systemic embolism, coronary artery injury, death
hyponatremia | periprocedural (at the time of the procedure and up to 1 month)
  serum sodium level < 135 mEq/L

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Natale, MD, Principal Investigator — Texas Cardiac Arrhythmia Institute, St. David's Medical Center
Locations (2):
- United States (2):
  - University of Colorado Hospital, Aurora, Colorado
  - Texas Cardiac Arrhythmia Institute, St. David's Medical Center, Austin, Texas